CLINICAL TRIAL: NCT06591910
Title: Induction Therapy With Serplulimab Combined With Chemotherapy Followed by Local Therapy for Unresectable Stage III Non-small Cell Lung Cancer
Brief Title: Induction Therapy With Serplulimab Combined With Chemotherapy for Unresectable Stage III Non-small Cell Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: LungMate-Unresectable
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Unresectable Stage III Non-small-cell Lung Cancer
Keywords: unresectable; stage III; non-small cell lung cancer; chemoimmunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative; Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Induction chemoimmunotherapy followed by surgery or radiotherapy for unresectable stage III NSCLC
  Interventions: Drug: Chemoimmunotherapy; Procedure: Surgery; Radiation: Radiation

INTERVENTIONS:
Drug: Chemoimmunotherapy — Induction Serplulimab combined with chemotherapy
Procedure: Surgery — After induction chemoimmunotherapy, patients with tumors resectable after chemoimmunotherapy will receive surgical treatment in department of thoracic surgery.
Radiation: Radiation — After induction chemoimmunotherapy, patients with tumors still unresectable will receive radiotherapy or other therapy.

SUMMARY:
For unresectable stage III (8th TNM) non-small cell lung cancer, chemoradiotherpay plus immunotherapy is recommended by PACIFIC trial. However, it is unclear whether induction chemoimmunotherapy followed by surgery or radiotherapy can provide good survival for this population. This prospective observational study aims to investigate the efficacy and safety of the therapeutic regimen of chemoimmunotherapy plus surgery/radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall sign the Informed Consent Form.
2. Aged 18 ≥ years.
3. Histological or cytological diagnosis of unresectable NSCLC by needle biopsy, and stage III (8th TNM) confirmed by imageological examinations (CT, PET-CT or EBUS).
4. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
5. Life expectancy is at least 12 weeks.
6. At least 1 measurable lesion according to RECIST 1.1.
7. Patients with good function of other main organs (liver, kidney, blood system, etc.)
8. Patients with normal lung function can tolerate surgery;
9. Without systematic metastasis (including M1a, M1b and M1c);
10. Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of Serplulimab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative.
11. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 days after chemotherapy or the last dose of Serplulimab (whichever is later).

Exclusion Criteria:

1. Participants who have received any systemic anti-cancer treatment for thymic epithelial tumor, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment;
2. Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;
3. With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment;
4. Participants who are allergic to the test drug or any auxiliary materials;
5. Participants with Interstitial lung disease currently;
6. Participants with active hepatitis B, hepatitis C or HIV;
7. Pregnant or lactating women;
8. Participants suffering from nervous system diseases or mental diseases that cannot cooperate;
9. Participated in another therapeutic clinical study;
10. Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresectable stage III (8th TNM) non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2030-09-20 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 60 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 6 months
  It refers to the proportion of patients who have had a complete response or partial response (according to RECIST1.1) as confirmed by CT evaluation after 3 weeks in all patients who have completed the neoadjuvant therapy. Only patients with measurable lesions at baseline will be analyzed.
Major pathologic response (MPR) | Up to 6 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery
Disease-free survival (DFS) | up to 60 months
  It refers to the time (months) from radical surgery to relapse or death of a participant due to disease progression. In the case of a patient who still survives at the time of analysis, the latest evaluation date will be used for interpolation (censoring).
Overall survival (OS) | up to 60 months
  It is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
R0 rate | Up to 6 months
  It is defined as the rate of complete resection with no residual tumor cell in the resection margin.
Severe adverse event (SAE) rate | up to 6 months
  It is defined as the frequency of severe adverse events from the participants enrolling to 30 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.
Health related quality of life (HRQol) | up to 6 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.

IPD SHARING:
Plan to Share IPD: Undecided